CLINICAL TRIAL: NCT04327375
Title: Effect of Body Composition on Thyroid Hormone Levels Among Overweight and Obese Subjects
Acronym: 3/2020
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Gianluigi Giannelli, Clinical Professor, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: 3/2020
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational: observational
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The study was aimed at investigating the relationship between body composition and thyroid hormone levels in overweight and obese subjects (BMI≥25 Kg/m2)

DETAILED DESCRIPTION:
Subjects were enrolled at the first examination whether they were not taking any medication, including oral contraceptives or drugs for osteoporosis, and free of significant medical illnesses, except obesity. Exclusion criteria were history of endocrinological diseases (diabetes mellitus, hypo or hyperthyroidism, hypopituitarism, etc.), chronic inflammatory diseases, stable known hypertension, angina pectoris, stroke, transient ischemic attack, heart infarction, congenital heart disease, malignancies, chronic inflammatory diseases, renal and liver failure, angina pectoris, myocardial infarction, heart failure, congenital heart diseases, minor and major stroke, and inherited thrombocytopenias and other major malignancies. Subjects were examined by means of the medical history, hormonal, metabolic and routine hematochemical parameters. The investigators provided for a clinical baseline evaluation that included extemporaneous ambulatory blood pressure (BP), bioimpedance and a physical assessment of body weight, Body Mass Index (BMI) and Waist Circumference (WC) as anthropometric parameters.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI> 25 Kg/m2)

Exclusion Criteria:

* Any kind of drug
* Hypertension
* Endocrine diseases (diabetes mellitus, hypo or hyperthyroidism, hypopituitarism, etc.),
* Chronic inflammatory diseases
* Renal failure
* Liver failure
* Angina pectoris
* Myocardial infarction and heart failure
* Genetic heart diseases
* Thrombocytopenias

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who came to the Outpatient Clinic of Nutrition at the National Institute of Gastroenterology "S. de Bellis," Research Hospital, Castellana Grotte, Italy.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Thyroid hormones (FT3, FT4) | Baseline
  FT3 (pg/mL), FT4 (pg/mL) concentration in serum
skeletal muscle mass | Baseline
  skeletal muscle mass (kg)
TSH | At baseline
  TSH (mU/L) concentration in serum

SECONDARY OUTCOMES:
Vitamin D | Baseline
  Vitamin D (ng/mL) concentration in serum
Insulin | Baseline
  Insulin (mIU/L) concentration in serum
eGFR (estimated glomerular filtration rate) | Baseline
  eGFR (ml/min/1.73 mq)
Creatinin | Baseline
  Creatinin (mg/dl) concentration in serum
Total cholesterol | Baseline
  Total cholesterol (mg/dL) concentrations in serum
HDL cholesterol | Baseline
  HDL cholesterol (mg/dL) concentrations in serum
LDL cholesterol | Baseline
  LDL cholesterol (mg/dL) concentrations in serum
BMI | Baseline
  BMI (kg/m^2)
Height | Baseline
  Height in meters
Weight | Baseline
  Weight in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Roberta Zupo, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zupo R, Castellana F, Sardone R, Lampignano L, Paradiso S, Giagulli VA, Triggiani V, Di Lorenzo L, Giannelli G, De Pergola G. Higher Muscle Mass Implies Increased Free-Thyroxine to Free-Triiodothyronine Ratio in Subjects With Overweight and Obesity. Front Endocrinol (Lausanne). 2020 Sep 29;11:565065. doi: 10.3389/fendo.2020.565065. eCollection 2020. PMID 33117281